CLINICAL TRIAL: NCT02172469
Title: A Comparison of 18 µg of Tiotropium Inhalation Capsules and Atrovent® Metered Dose Inhaler (2 Puffs of 20 µg, 4 Times Daily) in a Double-Blind, Double-Dummy, Efficacy and Safety Study in Adults With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety of Tiotropium and Atrovent in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.243
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium

ARMS (2):
- Tiotropium & Placebo (Experimental)
  Interventions: Drug: Tiotropium inhalation powder capsule; Drug: Placebo Metered Dose Inhaler
- Atrovent & Placebo (Active Comparator)
  Interventions: Drug: Ipratropium Bromide Metered Dose Inhaler; Drug: Placebo inhalation powder capsule

INTERVENTIONS:
Drug: Tiotropium inhalation powder capsule
  Arms: Tiotropium & Placebo
Drug: Placebo Metered Dose Inhaler
  Arms: Tiotropium & Placebo
Drug: Ipratropium Bromide Metered Dose Inhaler
  Other Names: Atrovent®
  Arms: Atrovent & Placebo
Drug: Placebo inhalation powder capsule
  Arms: Atrovent & Placebo

SUMMARY:
To compare the bronchodilator efficacy and safety of tiotropium inhalation capsules (18 µg once daily) and Atrovent® MDI (2 puffs of 20µg q.i.d.) among Filipino patients with COPD

ELIGIBILITY:
Inclusion Criteria:

* All patients had a diagnosis of chronic obstructive pulmonary disease according to the following criteria:

  * Patients had relatively stable airway obstruction with an FEV1 less than or equal to 65% of predicted normal and FEV1 less than or equal to 70% of FVC.
  * Predicted normal values were based on the guidelines for standardised lung function testing in the Philippines.
* Male or female patients 40 years of age or older.
* Patients had a smoking history of more than 10 pack-years. A pack-year is defined as the equivalent of smoking one pack of cigarettes per day for a year.
* Patients performed pulmonary function tests as required in the protocol.
* Patients were able to inhale medication from the Handihaler device and had a good technique of inhaling aerosol administered from an MDI.
* All patients signed an Informed Consent Form prior to participation in the trial i.e., prior to pre-study washout of their usual pulmonary medications.

Exclusion Criteria:

* Patients with significant diseases other than COPD were excluded. A significant disease was defined as a disease which in the opinion of the investigator could either put the patient at risk because of participation in the study or a disease which could influence the results of the study or the patient's ability to participate in the study.
* Patients with clinically significant abnormal baseline haematology, blood chemistry or urinalysis, if the abnormality defined a disease listed as an exclusion criterion, were excluded.
* All patients with a serum glutamate oxalacetate transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) twice the normal range, bilirubin 150% or creatinine 125% of the normal range were excluded regardless of the clinical condition. Repeated laboratory evaluations were not conducted in these subjects.
* Patients with a recent history (i.e. one year or less) of myocardial infarction were excluded.
* Patients with a recent history (i.e. three years or less) of heart failure or patients with any cardiac arrhythmia requiring drug therapy were excluded.
* Patients on regular use of daytime oxygen therapy were excluded.
* Patients with known active tuberculosis were excluded.
* Patients with a history of cancer within the last five years were excluded. Patients with treated basal cell carcinoma were allowed.
* Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis were excluded.
* Patients who have undergone pulmonary resection or a thoracotomy for any reason were excluded.
* Patients with an upper respiratory tract infection in the past 6 weeks prior to the screening visit (=visit 1) or during the baseline period of 2 weeks (run-in period) were excluded.
* Patients with known hypersensitivity to anticholinergic drugs, lactose or any other component of the inhalation capsule delivery system or the MDI were excluded.
* Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction were excluded.
* Patients with known narrow-angle glaucoma were excluded.
* Patients who were being treated with cromolyn sodium or nedocromil sodium were excluded.
* Patients who were being treated with antihistamines were excluded.
* Patients who were using oral corticosteroid medication at unstable (i.e. less than 6 weeks on a stable dose) or at a dose in excess of the equivalent 10 mg of prednisone per day or 20 mg every other day were excluded
* Pregnant or nursing women or women of childbearing potential who were not using a medically approved means of contraception (e.g. oral contraceptives, intrauterine devices, or diaphragm) were excluded.
* Patients with a history of asthma, allergic rhinitis or atopy or who had a blood total eosinophil count more or equal to 400 per μl (males) or more or equal to 320 per μl (females) were excluded. Repeated eosinophil counts were not conducted in these patients.
* Patients with a history and/or active alcohol or drug abuse were excluded.
* Patients who had taken an investigational drug one month or six half-lives (whichever is greater) prior to the screening visit (=visit 1) were excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2001-05; Primary Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in trough Forced Expiratory Volume in one second (FEV1) - Trough FEV1 response - | Baseline and week 4

SECONDARY OUTCOMES:
Through FEV1 response | week 2
FEV1 for the first 3 hours post drug administration on each pulmonary function test day | Day 1, 15 and 29
Trough Forced Vital Capacity (FVC) response | week 2 and 4
Individual FEV1 measurements | Day 1, 15 and 29
Individual FVC measurements | Day 1, 15 and 29
FVC for the first 3 hours post drug administration on each pulmonary function | Day 1, 15 and 29
Amount of salbutamol (MDI) use (rescue medication) | 4 weeks
Patient evaluation questionnaire (PEQ) | 4 weeks
PEFR (peak expiratory flow rate) measured by the patient | 4 weeks
Number of patients with adverse events | 4 weeks